CLINICAL TRIAL: NCT02131077
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind, Parallel-group, Phase I/II Clinical Study to Evaluate Safety and Efficacy of Allogeneic Adipose-derived Stem Cells for the Treatment of Lateral Epicondylitis
Brief Title: Safety and Efficacy Study of Allogeneic Adipose-derived Stem Cells for Treatment of Lateral Epicondylitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLO-ASC-TI-201
Record Dates: First submitted 2014-04-29; First posted 2014-05-06 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2014-05

CONDITIONS: Tennis Elbow
Keywords: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental): ALLO-ASC-TI injection
  Interventions: Biological: ALLO-ASC-TI
- Placebo (Placebo Comparator): Saline injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ALLO-ASC-TI
  Other Names: Allogenic adipose-derived stem cell
  Arms: treatment
Drug: Placebo
  Other Names: 0.9% Saline
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of allogeneic adipose-derived stem cells (ALLO-ASC) in patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 19 years.
2. Patients who are diagnosed as lateral epicondylitis (Pain≥4 of VAS during activity).
3. Patients who has sustained pain more than 6 months
4. Patients who lasting for pain in spite of conservative therapy
5. Patients who have one lesion under ultrasonic photography
6. Negative for urine beta-HCG for women of childbearing age
7. Patient who is able to give written informed consent prior to study start and to comply with the study requirements

Exclusion Criteria:

1. Patients who has been experienced steroid and prolotherapy or other treatment within 3 months at screening time
2. Patients who have lesion size of width and length more than 1 cm using ultrasonic photography test
3. Patients who were accompanied by the disease as follows: A. Arthritis of related joint to the target lesion (ex, cubital osteo- arthritis), B.Synovitis of related joint to the target lesion, C.Entrapment of related nerve to the target lesion(ex, radial tunnel syndrome), D.Generalized pain syndrome, E.Radiculopathy related to the target lesion(ex, cervical spodylosis ,cervical radicular syndrome), F.Rheumatoid arthritis, G.Previous fracture of arm causing limitations in arm function, H.Impaired sensibility, I.Paralysis
4. Patients who are pregnant or breast-feeding
5. Patients who have allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue
6. Patients who have history of fracture and dislocation at Ipsilateral upper extremity within 2 years recently
7. Patients who have operation history in tendon, ligament and bone at Ipsilateral upper extremity within 2 years recently
8. Patients who are unwilling to use an "effective" method of contraception during the study
9. Patients who have a clinically relevant history of abuse of alcohol or drugs
10. Patients who are considered not suitable for the study by investigator
11. Patients who have experienced treatment with stem cell before this study
12. Patients who currently enrolled in another investigational drug study within 30 days of screening

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | Week 12
  Improvement of VAS pain score at 12 weeks compared to baseline per each group

SECONDARY OUTCOMES:
VAS pain score | week 2, week 6 and week 12
  Changes in the VAS pain score during activity per each group
Improvement rate of VAS pain score | week 2, week 6 and week 12
  Improvement rate of VAS pain score at rest per each group
Modified Mayo Clinic Performance Index | week 2, week 6 and week 12
  Change in Modified Mayo Clinic Performance Index per each group
Ultrasonic photography | week 6 and week 12
  Change in analysis of lesion size per each group
Safety | Week 12
  Clinically measured abnormality of laboratory tests and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: S G Chung, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Asan Medical Center, Seoul
  - Chung-Ang University Hosptal, Seoul
  - Gangnam Severance Hospital, Seoul
  - Nanoori hospital, Seoul
  - Samsung medical center, Seoul
  - Seoul National University Hospital, Seoul